CLINICAL TRIAL: NCT01427868
Title: An Open-label, Phase I Study in Healthy Male Subjects to Compare the Pharmacokinetics of LB80331 and LB80317, Metabolites of LB80380, After a Single Oral Administration of LB80380 Free Base 150 mg (60 mg + 90 mg) Tablet or LB80380 Maleate Tablet 183 mg (150 mg as a Free Base)
Brief Title: Bioequivalence of LB80380 Free Base and Maleate Salt Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: LG-BVCL009
Record Dates: First submitted 2011-08-25; First posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Hepatitis B
Keywords: LB80380; bioequivalence
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LB80380 maleat salt (Experimental)
  Interventions: Drug: LB80380 maleate salt
- LB80380 free base (Active Comparator)
  Interventions: Drug: LB80380 free base

INTERVENTIONS:
Drug: LB80380 maleate salt — 183 mg (150 mg as a free base)
  Arms: LB80380 maleat salt
Drug: LB80380 free base — 150 mg
  Arms: LB80380 free base

SUMMARY:
The study is to compare pharmacokinetics of LB80331 and LB80317, which are the metabolites of LB80380, after a single oral administration of LB80380 free base 150 mg (60 mg + 90 mg) tablet or LB80380 maleate tablet 183 mg (150 mg as a free base) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male with good health
* 20 to 45 years of age at screening
* Body weight ±20% of ideal body weight
* Willingness and ability to comply with study procedures and communicate with investigators
* Provided written consent voluntarily after informed of all the pertinent aspects of the trial

Exclusion Criteria:

* Clinically significant abnormality on medical interview, physical examination, electrocardiogram or clinical laboratory evaluations
* Clinically significant acute or chronic medical conditions
* Use of prescriptive medicine within 14 days, or over-the-counter drug within 7 days before the first day of drug administration
* Participation in clinical trial within 3 months before the first day of drug administration
* Alcohol abuse
* Habitual smoker
* Habitual user of herbal medicine
* Use of grapefruit-containing food or grapefruit juice during the study period
* Positive drug abuse test and Positive HBs-antigen, HCV-antibody, or HIV-antibody test

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
AUC | up to 144 hours
Cmax | up to 144 hours

SECONDARY OUTCOMES:
Number of Participants with Adverse Events and Number of Adverse Events as a Measure of Safety and tolerability | up to 7 days
Profile of Pharmacokinetics | up to 144 hours
  Tmax, Aet, CL/F

CONTACTS AND LOCATIONS:
Overall Officials: Wooseong Huh, Prof, Principal Investigator — Samsung Medical Center
Locations (1):
- Clinical Trial Center, Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Jung JA, Kim SR, Kim TE, Kim JR, Lee SY, Huh W, Ko JW. Pharmacokinetic comparison of the maleate and free base formulations of LB80380, a novel nucleotide analog, in healthy male volunteers. Int J Clin Pharmacol Ther. 2012 Sep;50(9):657-64. doi: 10.5414/cp201716. PMID 22981147